CLINICAL TRIAL: NCT05347420
Title: Diagnostic Accuracy of Quantitative Neuropad Test for Diabetic Peripheral Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Rong Li, Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2020-403
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic peripheral neuropathy: Patients with diabetic peripheral neuropathy
  Interventions: Diagnostic Test: The visual Neuropad test and the quantitative Neuropad test
- non diabetic peripheral neuropathy: Patient without diabetic peripheral neuropathy
  Interventions: Diagnostic Test: The visual Neuropad test and the quantitative Neuropad test

INTERVENTIONS:
Diagnostic Test: The visual Neuropad test and the quantitative Neuropad test — The visual screening test includes whether the Neuropad test paper changes completely from blue to pink within 10 minutes (visual screening test a) and the time to complete color change (visual screening test b). the quantitative screening test using a handheld color scanner to scan the rate of color change, which estimated by the slope of the Neuropad color change per minute.

SUMMARY:
This study aimed to evaluate the diagnostic vaule of quantitative Neuropad for diabetic peripheral neuropathy

DETAILED DESCRIPTION:
This is a diagnostic study. Every patient will undertake Neuropad test, inculding the visual and quantitative screening tests. The visual screening test includes whether the Neuropad test paper changes completely from blue to pink within 10 minutes (visual screening test a) and the time to complete color change (visual screening test b). the quantitative screening test using a handheld color scanner to scan the rate of color change, which estimated by the slope of the Neuropad color change per minute. The visual and quantitative screening tests were compared when the Neuropathy Disability Score (NDS) and the Neurological Symptom Score (NSS) combined score as diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

1) diagnosed type 2 diabetic patients; 2) age between 18 and 80 years.

Exclusion Criteria:

1) patients with type 1 diabetes, secondary diabetes, and patients with pre-existing diabetic foot; 2) exclusion of the following clinical conditions: foot skin lesions (scarring, rash, flaking skin, infection, etc. on the skin of the test site), peripheral arterial occlusive disease, long-term heavy smoking, chronic alcohol abuse, thyroid disease, liver insufficiency (more than 3-fold increase in liver enzymes), renal insufficiency (eGFR ≤ 30 mL /min/1.73m2), acute and chronic infections, cervical and lumbar spine diseases, bone and joint system diseases, other neurological diseases, autoimmune diseases, malignant tumors, psychiatric or psychological diseases, taking drugs that affect autonomic function, and combined with other diseases that can cause peripheral neuropathy; 3) those who cannot complete the experiment as required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes in the inpatient ward of the Department of Endocrinology, The First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
The quantitative Neuropad test | 1 day
  The diagnostic vaule of quantitative Neuropad for diabetic peripheral neuropathy

SECONDARY OUTCOMES:
The visual Neuropad test | 1 day
  The diagnostic vaule of visual Neuropad for diabetic peripheral neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Rong Li, PHD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China